CLINICAL TRIAL: NCT06996093
Title: Chemotherapy Omission in Hormone Receptor(HR)-Positive/Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer With Lymph Node Negative Disease Receiving Adjuvant Endocrine Therapy and Cyclin-dependent Kinases 4 and 6 (CDK4/6) Inhibitor
Brief Title: Chemotherapy Omission in HR-positive/HER2-negative Breast Cancer With Lymph Node Negative Disease Receiving Adjuvant Endocrine Therapy and CDK4/6 Inhibitor
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor (MD, PhD), Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N087
Record Dates: First submitted 2025-04-30; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy omission; adjuvant ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Chemotherapy, Adjuvant; Aromatase Inhibitors

STUDY DESIGN:
Intervention Model Description: Arm #1: standard endocrine therapy plus CDK4/6 inhibitor without chemotherapy Arm #2: 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy, followed by standard endocrine therapy plus CDK4/6 inhibitor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm #1: Endocrine+CDK4/6i (Experimental): aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor without chemotherapy
  Interventions: Drug: aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor
- Arm #2: TC*4-Endocrine+CDK4/6i (Active Comparator): 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy, followed by aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor
  Interventions: Drug: 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy; Drug: aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor

INTERVENTIONS:
Drug: 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy — 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy
  Arms: Arm #2: TC*4-Endocrine+CDK4/6i
Drug: aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor — aromatase inhibitor (± ovarian suppression) plus CDK4/6 inhibitor

SUMMARY:
This is a prospective, randomized, open-label, multicenter phase III study to explore chemotherapy omission in hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancer with lymph node negative disease receiving adjuvant endocrine therapy and cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitor.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, multicenter phase III study to explore chemotherapy omission in hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancer with lymph node negative disease receiving adjuvant endocrine therapy and cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitor.

In this study, patient eligible will be randomized into either standard endocrine therapy plus CDK4/6 inhibitor without chemotherapy or standard endocrine therapy plus CDK4/6 inhibitor following 4 cycles of TC (docetaxel + cyclophosphamide) adjuvant chemotherapy.The safety and efficacy of each group will be assessed through invasive disease free survival (iDFS), disease-free survival (DFS), distant disease free survival (DDFS), overall survival (OS) and adverse effects (AE) as graded by Common Terminology Criteria for Adverse Events (CTCAE) 5.0 and patient reported outcome (PRO).

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged 18-70 years;
* ECOG performance status 0-1;
* Early-stage breast cancer, with postoperative pathology confirming invasive carcinoma, HR-positive and HER2-negative (In this study, HR-positive is defined as: ER-positive by IHC with >10% tumor cells staining positive; HER2-negative defined as HER2 0-1+ by IHC or HER2++ with negative FISH result, without amplification);
* Postoperative pathological stage pT2N0M0 and:

Histological grade 3, or Histological grade 2 with Ki67 ≥ 20% or high-risk multigene assay results;

* No prior neoadjuvant therapy received;
* Good postoperative recovery, with randomization occurring no more than 8 weeks after surgery;
* Normal function of major organs, meeting the following criteria:

Hematological tests must meet: HB ≥90 g/L (no transfusion within 14 days); ANC ≥1.5×10⁹/L; PLT ≥100×10⁹/L; Biochemical tests must meet: TBIL ≤1.5×ULN (upper limit of normal); ALT and AST ≤3×ULN; serum Cr ≤1.5×ULN;

* Contraception required for male participants and women of childbearing potential during treatment;
* Participants voluntarily enroll in the study, sign informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Bilateral breast cancer or carcinoma in situ (DCIS/LCIS);
* Metastasis at any site;
* Clinical or imaging suspicion of malignancy in the contralateral breast requiring biopsy (unless ruled out);
* Prior neoadjuvant therapy, including chemotherapy, radiotherapy, or endocrine therapy;
* Use of tamoxifen, raloxifene, or aromatase inhibitors (AIs) for breast cancer risk reduction ("chemoprevention") and/or osteoporosis treatment within the past 2 years;
* History of other malignancies within the past 5 years (except basal cell carcinoma of the skin or carcinoma in situ of the cervix), including contralateral breast cancer;
* Concurrent participation in another clinical trial;
* Severe systemic diseases and/or uncontrolled infections that preclude study participation;
* Severe cardiovascular or cerebrovascular events within 6 months before randomization (e.g., unstable angina, chronic heart failure, uncontrolled hypertension >150/90 mmHg, myocardial infarction, or stroke);
* Known hypersensitivity to the study drugs;
* Men and women of childbearing potential unwilling to use contraception during treatment and for 8 weeks after treatment completion;
* Pregnant or lactating women;
* Positive pregnancy test before study drug administration (for women of childbearing potential);
* Psychiatric disorders, cognitive impairment, or inability to comprehend the trial protocol, adverse effects, or comply with study procedures and follow-up (requires systematic evaluation before enrollment);
* Individuals lacking personal freedom or legal capacity for independent civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2508 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
invasive disease free survival | 4 years
  Invasive disease-free survival (IDFS), defined as occurrence of any of the following: ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer.

SECONDARY OUTCOMES:
distant disease free survival | 4 years
  Distant disease free survival refers to the proportion of people alive and without distant metastases at a specified period after diagnosis, even if they had a local recurrence
overall survival | 4 years
  Overall survival (OS), defined as the time from the start of the study to the occurrence of death.
adverse effects | 4 years
  adverse effects graded by Common Terminology Criteria for Adverse Events (CTCAE) 5.0
patient reported outcome | 4 years
  Information about a patient's health that comes directly from the patient. Examples of patient-reported outcomes include a patient's description of their symptoms, their satisfaction with care, and how a disease or treatment affects their physical, mental, emotional, spiritual, and social well-being. Lower scores in European Organization for Research and Treatment of Cancer(EORTC) QLQ-BR45 questionnaire will mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No